CLINICAL TRIAL: NCT01784887
Title: Clinical and Mechanistic Demonstration of a Bioelectric Dressing System for Non-healing Wound Management: A Phase II Randomized Trial
Brief Title: Clinical and Mechanistic Demonstration of a Bioelectric Dressing System for Non-healing Wound Management: A Phase II Trial
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Did not have study population to continue
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 370421; I-11-38 (Other Grant/Funding Number: AFMSA)
Record Dates: First submitted 2013-02-04; First posted 2013-02-06 (Estimated); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Non-healing Soft Tissue Wounds

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bioelectric Dressing (Active Comparator): SOC + Bioelectric Dressing
  Interventions: Drug: Procellera
- SOC (No Intervention): Standard of Care

INTERVENTIONS:
Drug: Procellera — PROCELLERA TM is an FDA-cleared bioelectrical dressing delivered in a sterile, single layer sheet consisting of a flexible polyester fabric layer containing silver and zinc, which are held in position on the polyester with a biocompatible binder.
  Other Names: Bioelectric Dressing
  Arms: Bioelectric Dressing

SUMMARY:
Utilizing wound healing trajectory analysis, patient-reported pain and QOL assessment, quantitative bacteriology, and inflammatory infiltrate quantification, an improvement in wound healing will be observed on a cellular, histomorphological and clinical level in the presence of a bioelectric dressing applied in conjunction with SOC.

DETAILED DESCRIPTION:
The PROCELLERA Antimicrobial Wound Dressing is considered a non-interactive wound dressing containing silver and zinc, classification product code MGP. Non-interactive wound dressings are considered by FDA to be non-significant risk, as per their Investigational Device Exemptions Manual (publication FDA 96-4159).

Procellera is FDA cleared under K081977 for professional use as a wound dressing for partial and full-thickness wounds.

Selection of Subjects

Type of the Subject Population

* At least 18 years old
* Male or female
* All ethnic groups

As a military-civilian cooperative Phase II prospective randomized trial, the study population will include chronic wound patients from both military and civilian backgrounds.

As incidence of complex non-healing wounds remains high in both military and civilian hospital settings, it is estimated that recruitment rate will be sufficiently rapid at each research site. While unanticipated delays (e.g. slow accrual) may occur, the limited patient population and length of time allotted for the clinical study (2 years) is assumed to offset any delays. A total of 60 participants will be enrolled studywide to obtain 50 evaluable participants from both sites combined. Up to 16 patients will be screened each day. A consecutive series of patients who meet the following inclusion/exclusion criteria and agree to participate will be recruited.

Inclusion and Exclusion Criteria

1. Inclusion Criteria > 18 years of age or older, male or female

   * Female subject not pregnant - pregnancy excluded by HCG (urine or serum) or by history (tubal ligation, hysterectomy, or menopause).
   * Have a non-healing external wound at any location of the body of ≥90 days duration that is (10-50 cm2) at initial screening and does not exceed 3 cm in depth.
   * May have a wound requiring Negative Pressure Wound Therapy in conjunction with standard of care wound treatment.
   * Subject is able to apply study dressing to his/her wound, or have a reliable and capable caregiver to do it.
   * Subjects will have adequate blood flow to the wound as defined by Skin Perfusion Pressure (SPP)47-49 of >30mmHg recorded over intact epidermis near the open wound margin.
   * Subjects with arterial repairs having adequate blood flow to the wound as defined by Skin Perfusion Pressure (SPP) of >30mmHg recorded over intact epidermis near the open wound margin.
   * Absence of clinical signs of infection (such as fever; malodorous wound exudate; increasing wound pain, drainage, erythema, friable granulation tissue and or edema).
   * Participant agrees to participate in follow-up evaluations.
   * Participant must be able to read and understand informed consent, and signs the informed consent.
2. Exclusion Criteria

   * Less than 18 years of age.
   * Pregnant or lactating woman.
   * Have undergone treatment with systemic corticosteroid or immunosuppressive therapy in the past 2 months.
   * Currently undergoing dialysis for renal failure.
   * Subject has wounds resulting from electrical burn, arterial insufficiency, chemical or radiation insult.
   * Subject has wounds with exposed bone, ligament, nerve, artery and/or tendon.
   * Active or previous (within 60 days prior to the study screening visit) chemotherapy.
   * Active or previous (within 60 days prior to the study screening visit) radiation to the affected wound area to be treated by study device or standard of care.
   * Physical or mental disability or geographical concerns (residence not within reasonable travel distance) that would hamper compliance with required study visits.
   * The Investigator believes that the subject will be unwilling or unable to comply with study protocol requirements, including application of bioelectric dressings, standard-of-care self-care requirements, and all study-related follow up visit requirements.
   * History of infection with Human Immunodeficiency Virus or other immunodeficiency disorders.
   * Heterotopic ossification underlying the wound based upon previous imaging or historical information from the subject's chart.
   * Severe anemia - Hgb < 7 g/dl (males) or < 6.5 (females) or coagulopathy (INR > 1.7).
   * Severe malnutrition (Albumin < 3.0 gm/dl; > 10% weight loss in preceding 6 weeks).
   * Allergy to silver or zinc.

ELIGIBILITY:
Inclusion Criteria:

> 18 years of age or older, male or female

* Female subject not pregnant - pregnancy excluded by HCG (urine or serum) or by history (tubal ligation, hysterectomy, or menopause).
* Have a non-healing external wound at any location of the body of ≥90 days duration that is (10-50 cm2) at initial screening and does not exceed 3 cm in depth.
* May have a wound requiring Negative Pressure Wound Therapy in conjunction with standard of care wound treatment.
* Subject is able to apply study dressing to his/her wound, or have a reliable and capable caregiver to do it.
* Subjects will have adequate blood flow to the wound as defined by Skin Perfusion Pressure (SPP)47-49 of >30mmHg recorded over intact epidermis near the open wound margin.
* Subjects with arterial repairs having adequate blood flow to the wound as defined by Skin Perfusion Pressure (SPP) of >30mmHg recorded over intact epidermis near the open wound margin.
* Absence of clinical signs of infection (such as fever; malodorous wound exudate; increasing wound pain, drainage, erythema, friable granulation tissue and or edema).
* Participant agrees to participate in follow-up evaluations.
* Participant must be able to read and understand informed consent, and signs the informed consent.

Exclusion Criteria:

* Less than 18 years of age.
* Pregnant or lactating woman.
* Have undergone treatment with systemic corticosteroid or immunosuppressive therapy in the past 2 months.
* Currently undergoing dialysis for renal failure.
* Subject has wounds resulting from electrical burn, arterial insufficiency, chemical or radiation insult.
* Subject has wounds with exposed bone, ligament, nerve, artery and/or tendon.
* Active or previous (within 60 days prior to the study screening visit) chemotherapy.
* Active or previous (within 60 days prior to the study screening visit) radiation to the affected wound area to be treated by study device or standard of care.
* Physical or mental disability or geographical concerns (residence not within reasonable travel distance) that would hamper compliance with required study visits.
* The Investigator believes that the subject will be unwilling or unable to comply with study protocol requirements, including application of bioelectric dressings, standard-of-care self-care requirements, and all study-related follow up visit requirements.
* History of infection with Human Immunodeficiency Virus or other immunodeficiency disorders.
* Heterotopic ossification underlying the wound based upon previous imaging or historical information from the subject's chart.
* Severe anemia - Hgb < 7 g/dl (males) or < 6.5 (females) or coagulopathy (INR > 1.7).
* Severe malnutrition (Albumin < 3.0 gm/dl; > 10% weight loss in preceding 6 weeks).
* Allergy to silver or zinc.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Clinical Efficacy | 2 years
  Assessment of the clinical efficacy of a bioelectric dressing in conjunction with standard-of-care on the healing rate of chronic soft tissue wounds compared with standard-of-care alone. In this 50-subject study, the primary endpoint for efficacy will be the rate of healing (healing trajectory) in the treatment group compared to that of the control group, during the 12-week treatment study period. It is hypothesized that a bioelectric dressing will reduce wound healing time when compared to SOC treatment, thereby accelerating wound healing trajectory.

SECONDARY OUTCOMES:
Dressing Efficacy | 2 Years
  To demonstrate the efficacy of a bioelectric dressing in the areas of enhanced and accelerated wound healing on a clinical, histomorphological and cellular level studied through wound healing with decreased incidence of bacterial infection, decreased pain levels for chronic non healing wounds studied through standard validated pain assessment tools, and improved quality of life (QOL), using complex non-healing wounds as a model for tissue response. Secondary endpoints for efficacy will be study wound inflammatory infiltrate, bacterial load, and patient reported pain and quality of life (QOL) by means of visual acuity score (VAS) and SF-12, respectively.

OTHER OUTCOMES:
No other outcome measures | No other outcome measures
  No other outcome measures

CONTACTS AND LOCATIONS:
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
no data

REFERENCES:
- [Background] Blount AL, Foster S, Rapp DA, Wilcox R. The use of bioelectric dressings in skin graft harvest sites: a prospective case series. J Burn Care Res. 2012 May-Jun;33(3):354-7. doi: 10.1097/BCR.0b013e31823356e4. PMID 21979844
- See also: Related Info — http://www.procellera.com/